CLINICAL TRIAL: NCT03989349
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Efficacy & Safety of Nemolizumab in Subjects With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.118169
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Moderate-to-Severe Atopic Dermatitis
Keywords: CD14152; Nemolizumab; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered via subcutaneous injection
  Interventions: Drug: Placebo
- Nemolizumab (Experimental): Nemolizumab administered via subcutaneous injection
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Nemolizumab — Nemolizumab
  Other Names: CD14152
  Arms: Nemolizumab

SUMMARY:
The main purpose of the study was to assess the efficacy and safety of nemolizumab after a 16-week treatment period in adult and adolescent subjects with moderate-to-severe atopic dermatitis (AD) not adequately controlled with topical treatments.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multi-center, parallel-group study in adult and adolescent subjects of age 12 years and above with moderate-to-severe AD. Eligible subjects had documented history of inadequate response to topical AD medication(s). Approximately 750 subjects were randomized in 2:1 to receive either nemolizumab or placebo, stratified by baseline disease severity (Investigator's Global Assessment (IGA) = 3, moderate; IGA = 4, severe) and peak pruritus numeric rating scale (PP NRS) severity (PP NRS >= 7; PP NRS < 7). A minimum of 250 subjects were randomized in each PP NRS strata. All nemolizumab-treated subjects who were clinical responders at Week 16 (i.e., the end of initial treatment [Initial Treatment Period]/beginning of Maintenance Period) were re-randomized (1:1:1) to different treatment regimens (nemolizumab injections Q4W or every 8 weeks (Q8W) [with placebo injections at Weeks 20, 28, 36, and 44 to maintain the blind] or placebo Q4W). A clinical responder was defined as a subject at Week 16 with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from baseline (EASI-75). All placebo-treated subjects who responded to placebo during the Initial Treatment Period continued to receive placebo Q4W in the Maintenance Period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged greater than and equal to (>=) 12 years at the screening visit.
* Chronic atopic dermatitis (according to American Academy of Dermatology Consensus Criteria) that has been present for at least 2 years before the screening visit.
* Eczema Area and Severity Index (EASI) score >=16 at the screening and baseline visits.
* Investigator Global Assessment (IGA) score >= 3 (scale of 0 to 4) at the screening and baseline visits.
* AD involvement >= 10 percent (%) of body surface area (BSA) at screening and baseline visits.
* Peak Pruritus Numerical Rating Scale (PPNRS) score of at least 4.0 at the screening and baseline visits.
* Documented recent history of inadequate response to topical medications (topical corticosteroids [TCS] with or without Topical calcineurin inhibitors [TCI]).
* Female subjects of childbearing potential (that is, fertile, following menarche and until becoming postmenopausal unless permanently sterile) must agree either to be strictly abstinent throughout the study and for 12 weeks after the last study drug injection or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.

Key Exclusion Criteria:

* Body weight (<) 30 kilograms (kg)
* Exacerbation of asthma requiring hospitalization in the preceding 12 months. Uncontrolled asthma in the preceding 3 months.
* Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 2 weeks before the baseline visit, or any confirmed or suspected coronavirus disease (COVID)-19 infection within 2 weeks before the screening or baseline visit.
* Pregnant women, breastfeeding women, or women planning a pregnancy during the clinical study.

Note: Subjects with chronic,stable use of prophylactic treatment for recurrent herpes viral infection can be included in this clinical study.

* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, e.g., monoclonal antibody) or to any of the study drug excipients.
* Any clinically significant issue, based on investigator judgement.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (138):
- United States (47):
  - Galderma Investigational Site 8749, Birmingham, Alabama
  - Galderma Investigational Site 8893, Birmingham, Alabama
  - Galderma Investigational Site 8866, Guntersville, Alabama
  - Galderma Investigational Site 8808, Scottsdale, Arizona
  - Galderma Investigational Site 8906, Bell Gardens, California
  - Galderma Investigational Site 8905, Canoga Park, California
  - Galderma Investigational Site 8577, Encinitas, California
  - Galderma Investigational Site 8673, Garden Grove, California
  - Galderma Investigational Site 8683, Los Angeles, California
  - Galderma Investigational Site 8907, Newport Beach, California
  - Galderma Investigational Site 8799, Ontario, California
  - Galderma Investigational Site 8745, Pasadena, California
  - Galderma Investigational Site 8658, San Diego, California
  - Galderma Investigational Site 8536, Santa Ana, California
  - Galderma Investigational Site 8820, Westminster, California
  - Galderma Investigational Site 8637, Farmington, Connecticut
  - Galderma Investigational Site 8875, Delray Beach, Florida
  - Galderma Investigational Site 8391, Hialeah, Florida
  - Galderma Investigational Site 8727, Hialeah, Florida
  - Galderma Investigational Site 8523, Largo, Florida
  - Galderma Investigational Site 8719, Miami, Florida
  - Galderma Investigational Site 8656, Miami, Florida
  - Galderma Investigational Site 8704, Miami, Florida
  - Galderma Investigational Site 8706, Miami, Florida
  - Galderma Investigational Site 8203, Tampa, Florida
  - Galderma Investigational Site 8839, Tampa, Florida
  - Galderma Investigational Site 8729, Rolling Meadows, Illinois
  - Galderma Investigational Site 8724, New Albany, Indiana
  - Galderma Investigational Site 8554, Detroit, Michigan
  - Galderma Investigational Site 8825, Las Vegas, Nevada
  - Galderma Investigational Site 8506, Hackensack, New Jersey
  - Galderma Investigational Site 8741, Buffalo, New York
  - Galderma Investigational Site 8723, Cortland, New York
  - Galderma Investigational Site 8733, New York, New York
  - Galderma Investigational Site 8823, Greensboro, North Carolina
  - Galderma Investigational Site 8030, Raleigh, North Carolina
  - Galderma Investigational Site 8747, Cincinnati, Ohio
  - Galderma Investigational Site 8212, Portland, Oregon
  - Galderma Investigational Site 8721, Pittsburgh, Pennsylvania
  - Galderma Investigational Site 8713, North Charleston, South Carolina
  - Galderma Investigational Site 8705, Chattanooga, Tennessee
  - Galderma Investigational Site 8807, Houston, Texas
  - Galderma Investigational Site 8618, Waco, Texas
  - Galderma Investigational Site 8003, Webster, Texas
  - Galderma Investigational Site 8672, Salt Lake City, Utah
  - Galderma Investigational Site 8896, Richmond, Virginia
  - Galderma Investigational Site 8434, Seattle, Washington
- Belgium (4):
  - Galderma Investigational Site 5448, Brussels
  - Galderma Investigational Site 6164, Ghent
  - Galderma Investigational Site 6038, Leuven
  - Galderma Investigational Site 6162, Liège
- Bulgaria (11):
  - Galderma Investigational Site 6029, Pleven
  - Galderma Investigational Site 6051, Sofia
  - Galderma Investigational Site 6078, Sofia
  - Galderma Investigational Site 6102, Sofia
  - Galderma Investigational Site 6165, Sofia
  - Galderma Investigational Site 6216, Sofia
  - Galderma Investigational Site 6046, Sofia
  - Galderma Investigational Site 6080, Sofia
  - Galderma Investigational Site 6079, Sofia
  - Galderma Investigational Site 6250, Sofia
  - Galderma Investigational Site 6251, Stara Zagora
- Estonia (3):
  - Galderma Investigational Site 6068, Tallinn
  - Galderma Investigational Site 6069, Tallinn
  - Galderma Investigational Site 6067, Tartu
- France (12):
  - Galderma Investigational Site 6198, Le Mans
  - Galderma Investigational Site 5031, Lille
  - Galderma Investigational Site 6170, Martigues
  - Galderma Investigational Site 6167, Nantes
  - Galderma Investigational Site 5140, Nice
  - Galderma Investigational Site 6133, Paris
  - Galderma Investigational Site 6166, Paris
  - Galderma Investigational Site 5407, Pierre-Bénite
  - Galderma Investigational Site 6135, Quimper
  - Galderma Investigational Site 6197, Toulon
  - Galderma Investigational Site 6169, Toulouse
  - Galderma Investigational Site 6168, Valence
- Georgia (8):
  - Galderma Investigational Site 6238, Tbilisi
  - Galderma Investigational Site 6227, Tbilisi
  - Galderma Investigational Site 6230, Tbilisi
  - Galderma Investigation Site 6228, Tbilisi
  - Galderma Investigational Site 6224, Tbilisi
  - Galderma Investigational Site 6235, Tbilisi
  - Galderma Investigational Site 6234, Tbilisi
  - Galderma Investigational Site 6236, Zugdidi
- Germany (16):
  - Galderma Investigational Site 5482, Aachen
  - Galderma Investigational Site 5566, Augsburg
  - Galderma Investigational Site 6082, Bonn
  - Galderma Investigational Site 6132, Dresden
  - Galderma Investigational Site 6031, Düsseldorf
  - Galderma Investigational Site 6083, Frankfurt
  - Galderma Investigational Site 5442, Gera
  - Galderma Investigational Site 6081, Goettigen
  - Galderma Investigational Site 6062, Halle
  - Galderma Investigational Site 6041, Hamburg
  - Galderma Investigational Site 6150, Hamburg
  - Galderma Investigational Site 6040, Hamburg
  - Galderma Investigational Site 5469, Heidelberg
  - Galderma Investigational Site 6086, Kiel
  - Galderma Investigational Site 6084, Mainz
  - Galderma Investigational Site 5382, Munich
- Hungary (6):
  - Galderma Investigational Site 6147, Budapest
  - Galderma Investigational Site 5513, Budapest
  - Galderma Investigational Site 5567, Debrecen
  - Galderma Investigational Site 6026, Debrecen
  - Galderma Investigational Site 6254, Gyula
  - Galderma Investigational Site 6053, Veszprém
- Italy (11):
  - Galderma Investigational Site 6145, Bologna
  - Galderma Investigational Site 6141, Chieti
  - Galderma Investigational Site 6045, L’Aquila
  - Galderma Investigational Site 6151, Parma
  - Galderma Investigational Site 6180, Pavia
  - Galderma Investigational Site 6143, Pisa
  - Galderma Investigational Site 6044, Roma
  - Galderma Investigational Site 6049, Roma
  - Galderma Investigational Site 6177, Rome
  - Galderma Investigational Site 6155, Rozzano
  - Galderma Investigational Site 6175, Vicenza
- Poland (17):
  - Galderma Investigational Site 5773, Bialystok
  - Galderma Investigational Site 6097, Chorzów
  - Galderma Investigational Site 5021, Katowice
  - Galderma Investigational Site 5362, Krakow
  - Galderma Investigational Site 6052, Krakow
  - Galderma Investigational Site 5363, Lodz
  - Galderma Investigational Site 5367, Lublin
  - Galderma Investigational Site 5377, Nowa Sól
  - Galderma Investigational Site 6063, Olsztyn
  - Galderma Investigational Site 6085, Poznan
  - Galderma Investigational Site 5495, Rzeszów
  - Galderma Investigational Site 6130, Szczecin
  - Galderma Investigational Site 6048, Tarnów
  - Galderma Investigational Site 6126, Warsaw
  - Galderma Investigational Site 5707, Warsaw
  - Galderma Investigational Site 6185, Wroclaw
  - Galderma Investigational Site 6096, Wroclaw
- Singapore (3):
  - Galderma Investigational Site 6124, Singapore
  - Galderma Investigational Site 6077, Singapore
  - Galderma Investigational Site 5499, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverberg JI, Rodriguez DN, Dias-Barbosa C, Filipenko D, Ulianov L, Piketty C, Puelles J. Psychometric Validation of the Subject Sleep Diary in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Apr;15(4):963-995. doi: 10.1007/s13555-025-01385-3. Epub 2025 Mar 21. PMID 40116983
- [Derived] Silverberg JI, Wollenberg A, Reich A, Thaci D, Legat FJ, Papp KA, Stein Gold L, Bouaziz JD, Pink AE, Carrascosa JM, Rewerska B, Szepietowski JC, Krasowska D, Havlickova B, Kalowska M, Magnolo N, Pauser S, Nami N, Sauder MB, Jain V, Padlewska K, Cheong SY, Fleuranceau Morel P, Ulianov L, Piketty C; ARCADIA 1 and ARCADIA 2 Study Investigators. Nemolizumab with concomitant topical therapy in adolescents and adults with moderate-to-severe atopic dermatitis (ARCADIA 1 and ARCADIA 2): results from two replicate, double-blind, randomised controlled phase 3 trials. Lancet. 2024 Aug 3;404(10451):445-460. doi: 10.1016/S0140-6736(24)01203-0. Epub 2024 Jul 24. PMID 39067461
- [Derived] Dias-Barbosa C, Silverberg JI, Stander S, Rodriguez D, Fofana F, Filipenko D, Ulianov L, Piketty C, Puelles J. Capturing patient-reported sleep disturbance in atopic dermatitis clinical trials. J Patient Rep Outcomes. 2024 Jul 15;8(1):73. doi: 10.1186/s41687-024-00751-7. PMID 39008191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 136 active sites in Belgium, Bulgaria, Estonia, France, Georgia, Germany, Hungary, Italy, Poland, Singapore, and the United States from 27 June 2019 to 26 September 2022.
Pre-assignment Details: A total of 787 randomized 2:1 to receive either nemolizumab or placebo.At Week 16, 235 nemolizumab treated participants were clinical responders(IGA of 0[clear] or 1[almost clear]or Eczema Area and Severity Index [EASI]-75) re-randomized to receive nemolizumab Q4,nemolizumab Q8W,or placebo during Maintenance Period.85 participants received placebo in Initial Treatment, responded to placebo at Week 16,re-assigned to placebo and continued to receive placebo Q4W in Maintenance Period.
Groups:
- Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg: Participants received nemolizumab 30 milligrams (mg) via 2 subcutaneous (SC) injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Initial Treatment Period (Baseline - Week 16 Predose): Placebo: Participants received placebo via 2 subcutaneous (SC) injections at Day 1, thereafter, every 4 weeks (Q4W) at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, every 8 weeks (Q8W) at Weeks 16, 24, 32, and 40 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W: Participants who received placebo, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
Period: Initial Treatment(Day 1-Week 16 Predose)
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W
Started | 522 | 265 | 0 | 0 | 0 | 0
Treated | 519 | 263 | 0 | 0 | 0 | 0
Safety Population (The safety population comprised all participants who received at least 1 dose of study drug.) | 519 | 263 | 0 | 0 | 0 | 0
Completed | 470 | 241 | 0 | 0 | 0 | 0
Not Completed | 52 | 24 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 24 | 15 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Physician/principal investigator decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not Treated | 3 | 2 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16-Week 48)
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16-Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16-Week 48): Placebo Q4W Re-assigned to Placebo Q4W
Started | 0 | 0 | 79 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 78 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 78 (Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders at Week 16 were re-randomized during Maintenance Period.) | 85 (Participants who received placebo, Q4W during Initial Treatment Period and were clinical responders at Week 16, were re-assigned during Maintenance Period.)
Treated | 0 | 0 | 78 | 78 | 77 | 84
Safety Population | 0 | 0 | 79 (One participant was re-randomized to Nemolizumab Q8W for Maintenance Period, but erroneously received Nemolizumb twice consecutively and thus counted in Nemolizumab 30 mg Q4W to Q4W for safety analysis.) | 77 | 77 | 84
Completed | 0 | 0 | 65 | 68 | 65 | 74
Not Completed | 0 | 0 | 14 | 10 | 13 | 11
Not completed — Lack of Efficacy | 0 | 0 | 2 | 2 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 4 | 2 | 2 | 0
Not completed — Re-randomized/Re-assigned but not Treated | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The ITT population consisted of all randomized participants.
Groups:
- Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg: Participants received nemolizumab 30 mg via 2 SC injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Initial Treatment Period (Baseline - Week 16 Predose): Placebo: Participants received placebo via 2 SC injections at Day 1, thereafter, Q4W at Weeks 4, 8, and 12 by a single SC injection during Initial Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Total
Number analyzed (Participants) | 522 | 265 | 787
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91 | 41 | 132
  Between 18 and 65 years | 394 | 209 | 603
  >=65 years | 37 | 15 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270 | 136 | 406
  Male | 252 | 129 | 381
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 19 | 63
  Not Hispanic or Latino | 464 | 244 | 708
  Unknown or Not Reported | 14 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 35 | 18 | 53
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 20 | 45
  White | 458 | 227 | 685
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Success at Week 16: Intent-To-Treat (ITT) Population
Description: IGA success was defined as an IGA score of 0 (clear) or 1 (almost clear) and at least a 2-grade improvement from baseline to Week 16. The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the Investigator or trained designee to evaluate the global severity of atopic dermatitis (AD) and the clinical response to treatment. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data at Week 16 were considered non-responders.
Time Frame: Week 16
Population: The ITT population consisted of all randomized participants. Data was planned to be collected and analyzed for Initial Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 37.7 | 26.0
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for the preceding outcome measure was statistically significant at two-sided 2.5% significance level; Test type: Other; p = 0.0006, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe] and PP NRS [>=7, <7]); Strata-adjusted percentage difference = 12.2, 97.5% CI 2-sided [4.6 to 19.8]

2. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Success at Week 16: Severe Pruritus Population
Description: IGA success was defined as an IGA score of 0 (clear) or 1 (almost clear) and at least a 2-grade improvement from baseline to Week 16. The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the Investigator or trained designee to evaluate the global severity of AD and the clinical response to treatment. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered a treatment failure. Participants with missing data at Week 16 were considered non-responders.
Time Frame: Week 16
Population: Severe pruritus population consisted of all randomized participants with a baseline PP NRS >=7. Data was planned to be collected and analyzed for Initial Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 36.7 | 22.0
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0008, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe]); Strata-adjusted percentage difference = 14.9, 97.5% CI 2-sided [5.6 to 24.3]

3. Primary Outcome: Percentage of Participants With >=75% Improvement in Eczema Area and Severity Index (EASI-75) at Week 16: ITT Population
Description: EASI-75 was defined as >=75 percent(%) improvement in EASI from baseline to Week 16. EASI evaluates severity of participants AD based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD(erythema, induration/papulation, excoriation and lichenification)scored separately for each of 4 body regions (head & neck, upper limbs, trunk & lower limbs on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI total score is composite score ranging from 0 to 72. Higher scores represent greater severity of AD. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered a treatment failure. Participants with missing data at Week 16 were considered non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 42.1 | 30.2
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 12.5, 97.5% CI 2-sided [4.6 to 20.3]

4. Primary Outcome: Percentage of Participants With >=75% Improvement in Eczema Area and Severity Index (EASI-75) at Week 16: Severe Pruritus Population
Description: as for outcome 3
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 41.1 | 25.0
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 16.3, 97.5% CI 2-sided [6.6 to 26.0]

5. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16: ITT Population
Description: The PP NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'. Weekly average PP NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 41.0 | 18.1
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for the preceding outcome measure was statistically significant at two-sided 2.5% significance level. Participants with missing data were considered non-responders; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 23.2, 97.5% CI 2-sided [16.1 to 30.3]
Statistical Analysis 2: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; Nemolizumab 30 mg versus Placebo using multiple imputation (MI) with missing at random (MAR) assumption; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 27.8, 97.5% CI 2-sided [21.2 to 34.5] — The estimates are from 50 complete datasets by MI-MAR assumption

6. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16: Severe Pruritus Population
Description: as for outcome 5
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 48.4 | 21.3
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting randomized stratification variables (IGA severity [3=moderate, 4=severe]; Strata-adjusted percentage difference = 27.1, 97.5% CI 2-sided [17.5 to 36.6]
Statistical Analysis 2: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; Nemolizumab 30 mg versus Placebo using MI-MAR assumption; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Strata-adjusted percentage difference = 33.4, 97.5% CI 2-sided [24.5 to 42.3] — The estimates are from 50 complete datasets by MI-MAR assumption

7. Secondary Outcome: Percentage of Participants With <2 Points in Weekly Average PP NRS at Week 16: ITT Population
Description: The PP NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'. Weekly average PP NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data were considered non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 28.4 | 11.3
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 17.1, 97.5% CI 2-sided [10.9 to 23.3]

8. Secondary Outcome: Percentage of Participants With <2 Points in Weekly Average PP NRS at Week 16: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 26.9 | 8.5
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 18.4, 97.5% CI 2-sided [11.0 to 25.8]

9. Secondary Outcome: Percentage of Participants With an Improvement of Sleep Disturbance Numeric Rating Scale (SD NRS) >=4 at Week 16: ITT Population
Description: The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants were asked the following question in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Weekly average SD NRS score was calculated using 7 consecutive days diary data and set to missing if less than 4 days data available. If a participant received any rescue therapy, the data after receipt of rescue therapy was considered treatment failure. Participants with missing data were considered non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 33.5 | 16.2
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 17.5, 97.5% CI 2-sided [10.8 to 24.3]

10. Secondary Outcome: Percentage of Participants With an Improvement of Sleep Disturbance Numeric Rating Scale (SD NRS) >=4 at Week 16: Severe Pruritus Population
Description: as for outcome 9
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 42.7 | 20.7
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 21.9, 97.5% CI 2-sided [12.5 to 31.4]

11. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 4: ITT Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 26.1 | 5.3
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — Strata-adjusted p-values were calculated from Cochran-Mantel-Haenszel test adjusting the randomized stratification variables (IGA severity and PP NRS); Strata-adjusted percentage difference = 20.9, 97.5% CI 2-sided [15.6 to 26.1]

12. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 4: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 30.4 | 7.9
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 22.5, 97.5% CI 2-sided [15.0 to 29.9]

13. Secondary Outcome: Percentage of Participants With Peak Pruritus Numeric Rating Scale (PP NRS) <2 at Week 4: ITT Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 15.9 | 2.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 13.2, 97.5% CI 2-sided [9 to 17.4]

14. Secondary Outcome: Percentage of Participants With Peak Pruritus Numeric Rating Scale (PP NRS) <2 at Week 4: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 11.1 | 1.2
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 9.9, 97.5% CI 2-sided [5.5 to 14.3]

15. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 2: ITT Population
Description: as for outcome 7
Time Frame: Week 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 16.9 | 1.9
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 15.1, 97.5% CI 2-sided [11 to 19.2]

16. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 2: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 19.3 | 3.0
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 16.3, 97.5% CI 2-sided [10.5 to 22.1]

17. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 1: ITT Population
Description: as for outcome 7
Time Frame: Week 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 522 | 265
percentage of participants | 6.7 | 0.4
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 6.4, 97.5% CI 2-sided [3.8 to 9.1]

18. Secondary Outcome: Percentage of Participants With Improvement of >=4 Points in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 1: Severe Pruritus Population
Description: as for outcome 7
Time Frame: Week 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo
Number analyzed (Participants) | 316 | 164
percentage of participants | 8.5 | 0.6
Statistical Analysis 1: Comparison: Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg vs Initial Treatment Period (Baseline - Week 16 Predose): Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was performed sequentially in order the outcome measures were reported and continued when the test for preceding outcome measure was statistically significant at two-sided 2.5% significance level; Test type: Other; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Strata-adjusted percentage difference = 8.0, 97.5% CI 2-sided [4.2 to 11.8]

ADVERSE EVENTS:
Time Frame: Initial Treatment Period: From baseline to Week 16 pre-dose; Maintenance Period: From end of Initial Treatment Period (i.e., Week 16) to Week 48
Description: The safety population comprised all participants who received at least 1 dose of study drug.
Groups:
- Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q8W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received nemolizumab 30 mg, every 8 weeks (Q8W) at Weeks 16, 24, 32, and 40 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W: Participants who received nemolizumab, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
- Maintenance Period (Week 16- Week 48): Placebo Q4W Re-assigned to Placebo Q4W: Participants who received placebo, Q4W during Initial Treatment Period and were clinical responders (defined as participants with an IGA of 0 (clear) or 1 (almost clear) or a >=75% improvement in EASI from Baseline) at Week 16 received placebo, Q4W at Weeks 16, 20, 24, 28, 32, 36, 40, and 44 by a single SC injection during Maintenance Period.
Arm/Group | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg | Initial Treatment Period (Baseline - Week 16 Predose): Placebo | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q4W | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q8W | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W | Maintenance Period (Week 16- Week 48): Placebo Q4W Re-assigned to Placebo Q4W
All-Cause Mortality (participants affected / at risk) | 0/519 | 0/263 | 0/79 | 0/77 | 0/77 | 0/84
Serious Adverse Events (participants affected / at risk) | 13/519 | 3/263 | 6/79 | 0/77 | 2/77 | 1/84
Other Adverse Events (participants affected / at risk) | 71/519 | 40/263 | 17/79 | 11/77 | 26/77 | 16/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg (N=519) | Initial Treatment Period (Baseline - Week 16 Predose): Placebo (N=263) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q4W (N=79) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q8W (N=77) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W (N=77) | Maintenance Period (Week 16- Week 48): Placebo Q4W Re-assigned to Placebo Q4W (N=84)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychogenic tremor (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period (Baseline - Week 16 Predose): Nemolizumab 30 mg (N=519) | Initial Treatment Period (Baseline - Week 16 Predose): Placebo (N=263) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q4W (N=79) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Q8W (N=77) | Maintenance Period (Week 16- Week 48): Nemolizumab 30 mg Q4W to Placebo Q4W (N=77) | Maintenance Period (Week 16- Week 48): Placebo Q4W Re-assigned to Placebo Q4W (N=84)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 34 (42) | 15 (15) | 6 (7) | 3 (4) | 6 (7) | 5 (5)
Nasopharyngitis (Infections and infestations) | 19 (24) | 12 (13) | 7 (12) | 3 (6) | 5 (6) | 6 (8)
COVID-19 (Infections and infestations) | 14 (14) | 8 (8) | 3 (3) | 4 (4) | 13 (13) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 5 (5) | 1 (1) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03989349/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT03989349/SAP_001.pdf